CLINICAL TRIAL: NCT04627298
Title: Normalizing Preteen HPV Vaccination With Practice-based Communication Strategies
Brief Title: Normalizing HPV Vaccination in Preteens With a Serious Video Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-1891; 1R01AI113305 (NIH)
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Human Papillomavirus
Keywords: vaccination; preteen; serious video game; human papillomavirus

STUDY DESIGN:
Intervention Model Description: Random assignment to intervention or comparison
Who Masked: Participant
Masking Description: On enrollment, participants randomly assigned to condition.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Game (Active Comparator): This arm tests use of video game to help preteens in the decision to pursue HPV vaccination. Participants in the intervention group are asked to play the Land of Secret Gardens game and complete 3 tasks: (1) play a shield game with blue spikey virus balls, (2) find hidden objects in 4 different garden sheds, and (3) create a potion (vaccine). Participants in the intervention arm are asked to respond to surveys about HPV and HPV vaccine knowledge, vaccination self-efficacy and decisional balance, the Physical/Emotional/Narrative Presence Scale (PENS) to gauge preteens' immersion in the game, and game play experience.
  Interventions: Behavioral: educational video game for preteens to support HPV vaccination
- No Video Game (No Intervention): This arm does not test the video game. Participants in the comparison arm are asked to respond to surveys about HPV and HPV vaccine knowledge, vaccination self-efficacy and decisional balance.

INTERVENTIONS:
Behavioral: educational video game for preteens to support HPV vaccination — An educational video game developed for 11-12 year olds to increase interest in and decision to pursue HPV vaccination.
  Arms: Video Game

SUMMARY:
Human papillomavirus (HPV) is the most common sexually transmitted infection in the United States and causes genital warts and cancers in both females and males. Vaccination against HPV is recommended for routine use in those aged 11-12 years old, yet is underutilized. The study's premise is that preteens are relevant decision makers who can be motivated to initiate and complete the HPV vaccine series (assuming parental consent and provider recommendation). This study evaluates a serious video game to engage preteens in the decision to pursue HPV vaccination. The hypothesis is that preteens who are assigned to the video game will be more likely to initiate and complete HPV vaccination than preteens who are not assigned to the video game.

DETAILED DESCRIPTION:
The aims of this pilot study are to (1) evaluate whether preteens who receive the video game have better self-reported outcomes related to knowledge of HPV and HPV vaccine, vaccination self-efficacy and decisional balance compared with preteens who do not receive the game; and (2) evaluate outcomes related to immersion in the video game and game play experiences of preteens who played the game. HPV vaccination initiation and completion data are collected from practices for both preteens who receive the game and a comparison group who do not receive the game.

This is a multiple baseline study based in primary care practices in North Carolina and conducted over 3 waves of 16 practices each wave. The goal is to recruit 160 boys and girls ages 11-12 and not vaccinated against HPV for each wave. Participants are recruited by their primary care providers to enroll in the study. Parents give consent and preteens give assent.

An original video game, Land of Secret Gardens, is created for the study. The game is a metaphor for protecting seedlings (body) with a potion (vaccine). Points to buy seeds and create the potion are earned by playing minigames. The minigames include several versions of finding secret objects in a garden shed and another involves playing a shield game with blue spikey balls (i.e., HPV) before they land on budding plants. Throughout the play, players are exposed to messaging about HPV and the benefits of the HPV vaccine.

Preteens are randomly assigned to an intervention group to play the video game or to a comparison group that will not play the game. Participants are asked to complete baseline and postintervention surveys. Measures included are scales for knowledge of HPV and HPV vaccine, vaccination self-efficacy and decisional balance about deciding to pursue HPV vaccination. Participants in the intervention group are also asked about story immersion and game play.

ELIGIBILITY:
Inclusion Criteria:

* preteens 11-12 who had not received any doses of HPV vaccination
* recruited by primary care practices in North Carolina
* parent signed HIPAA release
* willing to take baseline and postintervention surveys
* access to internet and mobile device or personal computer

Exclusion Criteria:

* preteens who had received at least one dose of HPV vaccine

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants Initiating vaccination with one dose of HPV vaccine | approximately 9 months post intervention for each cohort total
  HPV immunization records are obtained for all preteen participants from their primary care practices
Number of Participants completing HPV vaccination series with either 2 or 3 doses of HPV vaccine in accordance with vaccination schedule for participant | approximately 9 months post intervention for each cohort total
  HPV immunization records are obtained for all preteen participants from their primary care practices

SECONDARY OUTCOMES:
Mean HPV Vaccination Knowledge Scale Score (5 items, range 1-3) is collected from both intervention and comparison group participants via Qualtrics surveys; higher score indicates greater knowledge of HPV and HPV vaccination | Baseline and postintervention surveys 4 months apart
  Five items ask whether HPV vaccination can prevent genital warts, prevent cervical cancer, prevent anal cancer, prevent throat cancer, is recommended for 11-12 year old boys and girls
Mean HPV Vaccination Self-Efficacy Scale Score (8 items, range 1-3) is collected from both intervention and comparison group participants via Qualtrics surveys; higher score indicates greater confidence in getting HPV vaccination | Baseline and postintervention surveys 4 months apart
  Eight items ask how confident was participant in getting the HPV vaccine when consider side effects, pain, parental decision, faintness or dizziness, expense, inconvenience, weak recommendation from doctor, friends' knowledge of vaccination
Mean HPV Vaccination Decisional Balance Scale Score (4 items pro and 5 items con, range 1-3) is collected from intervention and comparison group participants via Qualtrics surveys; higher pro mean score and lower con mean score indicate greater support | Baseline and postintervention surveys 4 months apart
  Four items asked how important is the decision to get HPV vaccination (protection from HPV, protection from cancers and warts, protection from a sexually transmitted infection, and less likely to spread HPV); 5 items asked reasons for not getting HPV vaccination (too much time, too embarrassing to talk to parents, too embarrassing to talk to doctor, parents would not approve, parents would think participant was having sex)
Number of participants who evaluate video game characteristics via PENS: Physical/Emotional/Narrative Presence Scale (27 items) is collected from intervention group via Qualtrics; higher score indicates agreement with video game characteristic | Postintervention survey (4 months after completing baseline survey)
  Twenty seven items asked about participant immersion in the story: in-game autonomy, in-game competence, PENS questions related to immersion in the game, PENS questions related to intuitive controls, and interest and enjoyment
Number of participants who self-report characteristics of video game play (18 items) is collected from intervention group via Qualtrics; higher score indicates report of video game characteristic | Postintervention survey (4 months after completing baseline survey)
  Eighteen tasks are described in the video game, including playing a shield game with virus like balls, finding hidden objects in garden sheds, creating a vaccine potion

CONTACTS AND LOCATIONS:
Overall Officials: Bernard F. Fuemmeler, PhD, Study Director — Virginia Commonwealth University; Jamie L. Crandell, PhD, Study Director — University of North Carolina, Chapel Hill; Joan Cates, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Sandra J Diehl, MPH, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- Joan R, Cates, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cates JR, Fuemmeler BF, Diehl SJ, Stockton LL, Porter J, Ihekweazu C, Gurbani AS, Coyne-Beasley T. Developing a Serious Videogame for Preteens to Motivate HPV Vaccination Decision Making: Land of Secret Gardens. Games Health J. 2018 Feb;7(1):51-66. doi: 10.1089/g4h.2017.0002. Epub 2017 Nov 21. PMID 29161529
- [Derived] Cates JR, Fuemmeler BF, Stockton LL, Diehl SJ, Crandell JL, Coyne-Beasley T. Evaluation of a Serious Video Game to Facilitate Conversations About Human Papillomavirus Vaccination for Preteens: Pilot Randomized Controlled Trial. JMIR Serious Games. 2020 Dec 3;8(4):e16883. doi: 10.2196/16883. PMID 33270028